CLINICAL TRIAL: NCT04681391
Title: The Role of Implicit Attitude in the tDCS Modulation on Moral Decision-Making
Brief Title: tDCS, Moral Decision-Making, fMRI
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016B008
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Morality
Keywords: tDCS, Moral Decision-Making, Implicit Attitude, fMRI
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- anodal: For the active stimulation, which are anodal and cathodal tDCS, a constant current of 1 mA was delivered through 35 cm2 electrode for 20 minutes with fade-in and fade-out of 10 seconds, producing a current density of 0.029 mA/cm2. During anodal tDCS, the anode was placed over right temporoparietal junction, and the cathode was placed over left supraorbital area.
  Interventions: Device: transCranial direct current stimulation
- cathodal: For the active stimulation, which are anodal and cathodal tDCS, a constant current of 1 mA was delivered through 35 cm2 electrode for 20 minutes with fade-in and fade-out of 10 seconds, producing a current density of 0.029 mA/cm2. During cathodal tDCS, the cathode was placed over right temporoparietal junction, and the anode was placed over left supraorbital area.
  Interventions: Device: transCranial direct current stimulation
- sham (as a control condition): same fade-in, fade-out, and current density were applied for the sham stimulation, but the duration of current-delivering only last 35 seconds.
  Interventions: Device: transCranial direct current stimulation

INTERVENTIONS:
Device: transCranial direct current stimulation — In the present study, we applied DC Brain Stimulator Plus to stimulate right temporoparietal junction (rTPJ). The target electrode was placed over the location of rTPJ; on the other hand, the return electrode was placed over the left supraorbital area. That is, during anodal tDCS, the anode was placed over CP6, and the cathode was placed over left supraorbital area; conversely, during cathodal tDCS, the cathode was placed over CP6, and the anode was placed over left supraorbital area. For the active stimulation, which are anodal and cathodal tDCS, a constant current of 1 mA was delivered through 35 cm2 electrode for 20 minutes with fade-in and fade-out of 10 seconds, producing a current density of 0.029 mA/cm2. On the other hand, same fade-in, fade-out, and current density were applied for the sham stimulation, but the duration of current-delivering only last 35 seconds. Therefore, participants could feel the skin sensation but did not have the after-effects of tDCS.

SUMMARY:
Morality is the social rule about appropriateness of the behavior, containing concepts of justice, fairness, and rights. Previous studies suggested that the activation of right temporoparietal junction (rTPJ) should be involved in mental state reasoning in moral cognition. Implicit moral attitude, which reflects people's fundamental beliefs about right and wrong, could be assessed by implicit association test on moral scenarios (mIAT), as indicated by the D scores. According to our previous findings, we postulate that, during moral decision-making, the high D group would have less rTPJ involvement and the low D group would have more. Here we applied tDCS, a non-invasive neuromodulation technique, to modulate cortical excitability in rTPJ.

Based on our postulation, we divided participants into high D and low D group and hypothesized that tDCS over rTPJ would modulate the behavior depending on the group. The results revealed that, in aspect of mIAT, implicit moral attitude could be modulated differently depending on the group via tDCS over rTPJ. In addition, hemodynamic response within rTPJ showed a main effect of tDCS while carrying out the helping behavior. In conclusion, these findings indicated that tDCS over rTPJ could modulate the implicit moral attitude as well as the rTPJ activity during moral action.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers, are all ethnic Chinese, right-handed, and aged between 20 to 30 years old

Exclusion Criteria:

* any history of psychiatry or neurological disorders (e.g., dementia, seizures), head injury, and alcohol or substance abuse

Ages: 20 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Forty-two healthy volunteers (20 male; 22 female) without any history of psychiatry or neurological disorders (e.g., dementia, seizures), head injury, and alcohol or substance abuse, are all ethnic Chinese, right-handed, and aged between 20 to 30 years old (M = 23.476, SD = 2.211). They were recruited via the online survey sent to the student social group of National Yang-Ming University and National Taiwan University. Additionally, the study was approved by National Yang-Ming University Hospital, Yilan, Taiwan (IRB: 2016B008).
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Justice Sensitivity Inventory | 10 minutes
  Justice Sensitivity Inventory (JSI) is a self-report questionnaire which consists of four perspectives of justice sensitivity: victim, observer, beneficiary, and perpetrator (Schmitt, Baumert, Gollwitzer, & Maes, 2010; Schmitt, Gollwitzer, Maes, & Arbach, 2005). Each perspective contains ten descriptions, and participants would answer on a scale ranging from 1 (not at all) to 7 (exactly). Justice sensitivity reflects how people react to injustice and can be used to predict justice-related emotion and behavior (Baumert, Rothmund, Thomas, Gollwitzer, & Schmitt, 2013).
Morality Implicit Association Test | 15 minutes
  Implicit moral attitude was assessed by morality implicit association test (mIAT) in present study. The test was adapted from Implicit Association Test (IAT) developed by Greenwald and colleagues (1998). It measures the strength of the association 10 between target concepts and their associated attributes. In mIAT, target concepts were presented by morally good and morally bad clips, and attributes were presented by positive and negative words.
Moral Action Task | 10 minutes
  To verify the modulation of rTPJ activity via tDCS and to examine whether this modulation would alter people's moral behavior, participants would take the perspective of the active role while viewing moral scenarios in the MRI scanner.
  Forty-five dynamic visual stimuli from previous research were validated and applied in the Moral Action Task. Each animation consists of three still images with the respective duration of 1000ms, 200ms, and 200ms. These animations contain three kinds of moral scenarios: (1) a person who is taking an action to physically harm one another (perpetrating behavior); (2) a person who is alleviating the physical pain which the other one is suffered (helping behavior); and (3) a person who is carrying out an action that irrelevant to the other one (neural behavior). Additionally, the protagonists in these scenarios were all acting without the presence of faces, and therefore the participants would have no emotional clues for these social interactions.

SECONDARY OUTCOMES:
Moral Evaluation: Rating of Moral Action Task | 5 minutes
  Outside the MRI scanner, participants carried out the Moral Action Task again. They were instructed to imagine themselves as the actor in the animation and pressed the button just like they really did the moral actions. Moreover, they were asked how much guilt or warm-glow after doing the action. The ratings were on a visual analog scale ranging from 1 to 7 points (Yoder & Decety, 2014).

REFERENCES:
- [Background] Ciaramelli E, Muccioli M, Ladavas E, di Pellegrino G. Selective deficit in personal moral judgment following damage to ventromedial prefrontal cortex. Soc Cogn Affect Neurosci. 2007 Jun;2(2):84-92. doi: 10.1093/scan/nsm001. PMID 18985127
- [Background] FeldmanHall O, Mobbs D, Evans D, Hiscox L, Navrady L, Dalgleish T. What we say and what we do: the relationship between real and hypothetical moral choices. Cognition. 2012 Jun;123(3):434-41. doi: 10.1016/j.cognition.2012.02.001. Epub 2012 Mar 9. PMID 22405924
- [Background] Fumagalli M, Priori A. Functional and clinical neuroanatomy of morality. Brain. 2012 Jul;135(Pt 7):2006-21. doi: 10.1093/brain/awr334. Epub 2012 Feb 13. PMID 22334584
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Result] Gaesser B, Hirschfeld-Kroen J, Wasserman EA, Horn M, Young L. A role for the medial temporal lobe subsystem in guiding prosociality: the effect of episodic processes on willingness to help others. Soc Cogn Affect Neurosci. 2019 May 17;14(4):397-410. doi: 10.1093/scan/nsz014. PMID 30809675
- [Result] Santiesteban I, Banissy MJ, Catmur C, Bird G. Enhancing social ability by stimulating right temporoparietal junction. Curr Biol. 2012 Dec 4;22(23):2274-7. doi: 10.1016/j.cub.2012.10.018. Epub 2012 Nov 1. PMID 23122848